CLINICAL TRIAL: NCT04475770
Title: Effect of Sustained Natural Apophyseal Glides on Stiffness of Lumbar Stabilizer Muscles in Non-specific Low Back Pain Individuals
Brief Title: Effect of SNAGs on Stiffness of Lumbar Stabilizer Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yunus Emre Tutuneken, Research assistant, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Low Back Pain; Manuel Therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real SNAGs (Experimental): Real SNAGs group consists of 16 participants, where the Mulligan concept lumbal SNAGs is applied and evaluations are made before and after.
  Interventions: Other: Real Sustained Natural Apophyseal Glides (SNAGS)
- Sham SNAGs (Sham Comparator): The Sham SNAGs group consists of 16 participants who performed the same positioning as the Real SNAGs group and evaluated twice with a similar interval without any intervention to the spine.
  Interventions: Other: Sham Sustained Natural Apophyseal Glides (SNAGS)

INTERVENTIONS:
Other: Real Sustained Natural Apophyseal Glides (SNAGS) — Manual therapists use treatment modalities that include passive techniques such as mobilization and manipulation. Mobilization with movement (MWM) developed by Mulligan involves applying a sustained transverse glide to the spinous process of a vertebra while actively or passively performing. These techniques have gained the name "Sustained Natural Apophyseal Glides" (SNAGS) as it is maintained at the pain-free range and follows the plane of the apophyseal joints under treatment.
  Arms: Real SNAGs
Other: Sham Sustained Natural Apophyseal Glides (SNAGS) — The participants in the Sham SNAGs group will be positioned same as the SNAG group. Mulligan belt will be used, which included the patient's waist and physiotherapist's hip. The physiotherapist will place the hypothenar region of his hand on the spinous processes of the symptomatic lumbar spine levels and waited a few seconds without no glide will be performed. Sham SNAGs practice consisted of 3 sets of 6 repetitions and a 60-second rest period was given between the sets.
  Arms: Sham SNAGs

SUMMARY:
Low back pain is a common health problem worldwide. Epidemiological studies have shown that 70-80% of all people are affected at least once in their lifetime. Although it is common, often the cause of the pain has not been determined and is called 'nonspecific low back pain.

Low back pain has been shown to alter the structure of deep and superficial muscles such as multifidus and erector spinae. However, it has not been fully explained how changes in muscle fiber structure affect the biomechanical properties and functions of the muscle.

There are various manual therapy techniques in the treatment of low back pain. Manual therapists use treatment modalities that include passive techniques such as mobilization and manipulation. Mobilization with movement (MWM) developed by Mulligan involves applying a sustained transverse glide to the spinous process of a vertebra while actively or passively performing. These techniques have gained the name "Sustained Natural Apophyseal Glides" (SNAGS) as it is maintained at the pain-free range and follows the plane of the apophyseal joints under treatment.

Ultrasound shear wave elastography (SWE) provides an advantage since it can quantitatively assess tissue elasticity of in vivo skeletal muscles through non-invasive high-frequency ultrasound waves.

The aim of this study was to investigate the acute effect of Mulligan SNAGs on the stiffness of muscle tissue by using Ultrasound shear wave elastography which is an objective assessment technique.

ELIGIBILITY:
Inclusion Criteria:

* patients who diagnosed with non-specific low back pain
* between the ages of 18-24
* patients who able to perform at least 40° of trunk flexion

Exclusion Criteria:

* patients who obese, pregnant, had specific low back pain
* indication for surgery in the past 1 year
* the trauma of lumbar region, and systemic inflammatory disease affecting this area
* exercise and conventional physiotherapy in the last 6 months

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
muscle stiffness | 4 weeks
  The muscle stiffness of lumbar back muscles will be assessed using the B-mode of the ultrasound Shear Wave Elastography (SWE) imaging device. Longitudinal ultrasound Shear Wave Elastography images of the multifidus and erector spinal muscles will be taken bilaterally with a linear array probe in the prone position.

SECONDARY OUTCOMES:
The sit and reach test | 4 weeks
  The sit and reach test will be used for back and leg flexibility.
Visual Analogue Scale | 4 weeks
  Pain will be measured with Visual Analogue Scale. Visual Analogue Scale is the most commonly used method for measuring the pain level.
  It is scored between 0 and 10. 0 means no pain (minimum score) 10 means I have unbearable pain (maximum score). Higher score means worse result.
The Functional Reach Test | 4 weeks
  The Functional Reach Test will be used to measure standing balance. While the contact surface of the person was in contact with the ground, the distance between the length of the arm and its maximum reach will be measured.
The Flamingo Balance Test | 4 weeks
  The Flamingo Balance Test is total body balance test, and forms part of the Eurofit Testing Battery. This single leg balance test assesses the strength of the leg, pelvic, and trunk muscle as well as dynamic balance. purpose: To assess the ability to balance successfully on a single leg.
Lateral bridge test | 4 weeks
  side-bridge test, assesses muscular endurance of the lateral core muscles (i.e., transverse abdominis, obliques, quadratus lumborum, and erector spinae). Similar to the trunk flexor endurance test, this timed test involves static, isometric contractions of the lateral muscles on each side of the trunk that stabilize the spine.
Trunk extensor endurance | 4 weeks
  The trunk extensor endurance test is generally used to assess muscular endurance of the torso extensor muscles (i.e., erector spinae, longissimus, iliocostalis, and multifidi). This is a timed test involving a static, isometric contraction of the trunk extensor muscles that stabilize the spine.
The Oswestry Disability Index | 4 weeks
  The functional level will be assessed using The Oswestry Disability Index (ODI) that ıs consist of 10-item. These items assessed pain intensity, personal care, lifting, walking, sitting, sleeping, sex life, and social life. Each item is numbered between from 0 to 5. As the total score increases, the level of disability increases. Each item is number between 0 to 5. As the total score increases, the level of disability increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No